CLINICAL TRIAL: NCT04795050
Title: Mitigating Cardiovascular Disease Risk Among Rural Diabetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Laurie Abbott, Assistant Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC # 2018 23127
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Health Promotion

STUDY DESIGN:
Intervention Model Description: Cluster randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Project POWER
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Project POWER — Diabetes health promotion/cardiovascular disease risk reduction educational curriculum
  Arms: Intervention

SUMMARY:
The study explored the effects of the cardiovascular disease risk reduction intervention on diabetes fatalism, self-care activities, social support, knowledge, perceived self-managment among a rural population.

DETAILED DESCRIPTION:
An experimental pretest-posttest control group design was used to assess the effects of a diabetes health promotion intervention among participants recruited from rural churches located in the southern United States. The intervention, called Project Power, is a culturally relevant, church-based diabetes education program that was developed by the American Diabetes Association (ADA). Participating churches were randomized to experimental and control groups using random numbers tables having numerical parity no greater than 2. Since an individual church is the unit of randomization, all of the participants in that church received the same treatment condition. Churches randomized to the intervention group received the health promotion program, and those designated to the control group received an educational brochure. Recruitment, data collection and intervention delivery, for the intervention group, occurred on the church grounds.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified African Americans aged 22 years or older, who have been diagnosed with Diabetes Mellitus, Type 1 or 2

Exclusion Criteria:

* Other than African American, younger than 22 years of age

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Diabetes Self-care Activities | Baseline
  The Summary of Diabetes Self-care Activities (SDSCA) (Toobert, Hampson, & Glascow, 2000) includes multiple choice questions and items about self-care behaviors answered in days per week. The internal consistency of the instrument is adequate (α = .71). The scores ranged from a minimum of 0 to a maximum of 105. Higher scores indicated better diabetes self-care.
Diabetes Knowledge | Baseline
  The Revised Diabetes Knowledge Test: Michigan Diabetes Research Center (Fitzgerald et al., 2016) is a 23-item multiple choice diabetes knowledge test. The scale has good reliability for both the general test (α = .77) and the insulin use subscale (α = .84). The twenty scored items were worth 5 points each for a maximum of 100 points total. Higher scores indicated higher knowledge levels.
Change from Baseline Diabetes Self-care Activities at Three Weeks | Three weeks after baseline
  The Summary of Diabetes Self-care Activities (SDSCA) (Toobert, Hampson, & Glascow, 2000) includes multiple choice questions and items about self-care behaviors answered in days per week. The internal consistency of the instrument is adequate (α = .71). The scores ranged from a minimum of 0 to a maximum of 105. Higher scores indicated better diabetes self-care.
Change from Baseline Diabetes Knowledge at Three Weeks | Three weeks after baseline
  The Revised Diabetes Knowledge Test: Michigan Diabetes Research Center (Fitzgerald et al., 2016) is a 23-item multiple choice diabetes knowledge test. The scale has good reliability for both the general test (α = .77) and the insulin use subscale (α = .84). The twenty scored items were worth 5 points each for a maximum of 100 points total. Higher scores indicated higher knowledge levels.

SECONDARY OUTCOMES:
Diabetes Fatalism | Baseline and three weeks later
  The Diabetes Fatalism Scale (Egede & Ellis, 2010) is a 12-item, 6-point Likert scale that measures the three constructs associated with diabetes fatalism: emotional distress, coping, and self-efficacy. The measure has excellent internal consistency (α = .83). The total score ranged from a minimum of 12 points and maximum of 72 points. Higher scores indicated greater diabetes fatalism.
Perceived Diabetes Self-Management | Baseline and three weeks later
  The Perceived Diabetes Self-Management Scale (PDSMS) (Wallston, Rothman, & Cherrington, 2007) is an 8-item, Likert scale-type tool with responses that range from "Strongly Disagree" (1) to "Strongly Agree" (5) for each of the 8 items. The tool measures self-care perceptions and has excellent internal consistency (α = .83). The total score ranged from a minimum of 8 points and maximum of 40. Higher scores indicate greater perceptions of diabetes self-management.
Social Support | Baseline and three weeks later
  The Medical Outcomes Study Social Support Survey (Sherbourne & Stewart, 1991) is a instrument that has one fill-in-the-blank and 19 Likert scale, 5-point items that range from "None of the Time" (1) to "All of the Time" (5). The four social support subscales have excellent reliabilities (α = .91 - .97). The possibility of ranges were between 19 and 95, and higher scores indicated higher social support.
Change from Baseline Diabetes Fatalism at Three Weeks | Baseline and three weeks later
  The Diabetes Fatalism Scale (Egede & Ellis, 2010) is a 12-item, 6-point Likert scale that measures the three constructs associated with diabetes fatalism: emotional distress, coping, and self-efficacy. The measure has excellent internal consistency (α = .83). The total score ranged from a minimum of 12 points and maximum of 72 points. Higher scores indicated greater diabetes fatalism.
Change from Baseline Perceived Diabetes Self-Management at Three Weeks | Baseline and three weeks later
  The Perceived Diabetes Self-Management Scale (PDSMS) (Wallston, Rothman, & Cherrington, 2007) is an 8-item, Likert scale-type tool with responses that range from "Strongly Disagree" (1) to "Strongly Agree" (5) for each of the 8 items. The tool measures self-care perceptions and has excellent internal consistency (α = .83). The total score ranged from a minimum of 8 points and maximum of 40. Higher scores indicate greater perceptions of diabetes self-management.
Change from Baseline Social Support at Three Weeks | Baseline and three weeks later
  The Medical Outcomes Study Social Support Survey (Sherbourne & Stewart, 1991) is a instrument that has one fill-in-the-blank and 19 Likert scale, 5-point items that range from "None of the Time" (1) to "All of the Time" (5). The four social support subscales have excellent reliabilities (α = .91 - .97). The possibility of ranges were between 19 and 95, and higher scores indicated higher social support.

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University College of Nursing, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No